CLINICAL TRIAL: NCT04045249
Title: Comparison Between Different Feeding Protocols and Existing Protocol for the Treatment of Acute Malnutrition (A Cluster Randomized Controlled Clinical Trial)
Brief Title: Comparison of Different Feeding Protocols for the Treatment of Acute Malnutrition
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Integrated Reproductive Maternal Newborn & Child Health and Nutrition Program, Punjab (Other Government)
Responsible Party: Principal Investigator, Dr. Zahra Khan, Principal Investigator, Integrated Reproductive Maternal Newborn & Child Health and Nutrition Program, Punjab
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: RUTF18
Record Dates: First submitted 2019-07-29; First posted 2019-08-05 (Actual); Last update posted 2019-08-05 (Actual); Status verified 2019-08

CONDITIONS: Malnutrition, Child
Keywords: Malnutrition; RUTF; Children; Home base food
MeSH Terms: conditions — Child Nutrition Disorders; Malnutrition

STUDY DESIGN:
Intervention Model Description: Study involved 3 arms; 1st arm was treated as per standard protocol. 2nd arm was provided half calories from RUTF and half from home based food, 3rd arm was provided home based food along with MMS
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- 1st Group (No Intervention): Children were treated as per standard CMAM protocols; provided RUTF until MUAC reaches 11.5 cm
- 2nd Group (1st Intervention group) (Experimental): Children were initially provided RUTF until MUAC reach 11 cm then 50 % calories were provided from RUTF and 50% calories from home based food
  Interventions: Dietary Supplement: Home based food
- 3rd Group (2nd Intervention) (Experimental): Children were initially provided RUTF until MUAC reach 11 cm then 100 % calories provided from home based food
  Interventions: Dietary Supplement: Home based food

INTERVENTIONS:
Dietary Supplement: Home based food — Home based food is compare able to RUTF
  Arms: 2nd Group (1st Intervention group); 3rd Group (2nd Intervention)

SUMMARY:
Though malnutrition is prevalent worldwide but its situation is alarming in low- and middle-income countries. Pakistan has also been facing an alarming situation of prevailing severe malnutrition. Malnutrition in its any form costs a huge intolerable burden not only on national health care system, but also on social and economic fabric of the nation. The current management of severe malnutrition is based on World Health Organization (WHO) guidelines and protocols which has been evolved from expert opinions and observational studies. The principles of these protocols have emerged from emergency settings and converting these protocols for developing countries where severe malnutrition, a routine burden is a critical challenge. In the absence of standard protocols for the treatment of uncomplicated severe malnutrition in non-emergency settings it is important to test and optimize different approaches to treat severely acute malnutrition (SAM). It is hypothesized that by optimizing, adapting and implementing time oriented and resource intensive approaches, a huge burden of high cost of RUTF may be reduced. While RUTF may be utilized to treat SAM children in emergency settings, it is not a substitute of local household foods. Therefore, a pilot study has been conducted to compare the various treatment protocols for malnourished children. We specifically hypothesized that a reduced dose of RUTF for reduced duration, combined with age-appropriate food intake from locally available resources can treat uncomplicated SAM children cost effectively as compared to standard national Community Management of Acute Malnutrition (CMAM) protocol currently implemented in Punjab, Pakistan.

DETAILED DESCRIPTION:
Malnutrition signifies to inadequacies, immoderations or imbalances in an individual's consumption of nutrients or energy. The word malnutrition covers both under and over-nutrition. Undernutrition manifest in two different ways acute and chronic malnutrition. The acute malnutrition includes wasting while chronic malnutrition includes stunting. The situation of malnutrition has been perplexed in Pakistan in recent years and according to National Nutrition Survey (2018) rates of wasting are alarmingly high. Also, Pakistan ranks at 2nd position for infant and child mortality. The standard treatment of uncomplicated SAM in Pakistan often utilizes prolonged use of therapeutic food (RUTF), and after discharge results in high rates of relapse(official data from department of Health doesn't support this statement, according to them there is low rate of relapse). The present pilot study was conducted with the objective to find cost effective treatment protocols for treatment of uncomplicated SAM children. The study was conducted at The Children's Hospital and Institute of Child Health, Lahore in Out Patient Therapeutic Program (OTP) of Preventive Pediatrics Department. The children diagnosed with SAM aged 6-59 months without any specific gender preference were recruited. Weight, height and MUAC were measured at the time of enrolment in the study and Weight for Height (WHZ), Weight for Age (WAZ), Height for Age (HAZ) standard deviation (SD) Z scores and weight velocity was calculated for baseline. For current pilot study SAM children were grouped into 3 clusters. First, 30 children were grouped in 1st cluster, next 30 in 2nd cluster and further next 30 in 3rd cluster. Children in 1st cluster were treated as per standard CMAM protocols. Children in this cluster were provided RUTF as per admission weight of child until they attain 11.5cm MUAC or >-3SD WHZ. The children in the 2nd group (1st intervention group) were initially provided RUTF until they attain MUAC 11cm. After this, children were provided 50% of their required daily calories intake by RUTF and 50% of the calories were provided by the home-based food. The children in the 3rd group (2nd intervention group) were initially provided RUTF until they attain MUAC 11 cm. After this, children were provided their 100% caloric requirement from home-based food along with micronutrients sachets (MMS). The discharge criteria for control group was according to the existing CMAM guidelines that is MUAC > 11.5 cm. The discharge criteria for 2nd & 3rd group was MUAC > 12.5 cm and WHZ > -2SD score. Follow-up home visits of all children were done according to a predefined protocol. During follow-up the control and intervention groups underwent weekly anthropometric measurements. Follow up of the study participants of each group was continued for one month. Growth rate, recovery rate, mortality rate, relapse frequency and duration of recovery were calculated for each group.

ELIGIBILITY:
Inclusion Criteria:

* Children 6-59 months with MUAC <11.5cm and Weight for Height Z score < -3SD
* Having good appetite, alert and clinically well

Exclusion Criteria:

* WHZ score - 4 SD
* MUAC < 8 cm
* Secondary malnutrition diagnosed by a gastroenterologist and dietitian
* Family History
* Birth Anomolies
* Any hidden/ asymptomatic health conditions
* Any patient coming from out of city (Lahore)
* Anorexia
* High fever (>104 F)
* Severe pallor
* Severe dehydration
* Lower respiratory tract infection
* Bipedal edema
* Visible severe wasting

Ages: 6 Months to 59 Months | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 90 (Actual)
Dates: Start 2018-12-10 (Actual); Primary Completion 2019-04-25 (Actual); Study Completion 2019-04-25 (Actual)

PRIMARY OUTCOMES:
Growth velocity | 3 months
  Weight in Kg
Growth velocity | 3 months
  Height in cm
Growth velocity | 3 months
  Mid Upper Arm Circumference (MUAC) in cm
Duration of recovery from SAM | 3 months
  Time required each child to reach MUAC > 11.5
Rate of relapse | 3 months
  Number of children relapsed during the trial
Rate of mortality | 3 months
  Number of children dying during trial

SECONDARY OUTCOMES:
Rate of recovery from Moderate Acute Malnutrition in 1st group | 3 months
  Proportion of children who reach MUAC > 12.5 cm
Number of children having diarrhoea and acute respiratory infection during trial | 3 months
Number of children not coming for follow up visits due to any reason | 3 months

CONTACTS AND LOCATIONS:
Overall Officials: Zahra Khan, PhD, Principal Investigator — IRMNCH & Nutrition Program
Locations (1):
- The Children's Hospital & The Institute of Child Health, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No